CLINICAL TRIAL: NCT07021976
Title: A Multicentre, Randomized, Double-blind, Placebo-parallel-controlled Phase III Clinical Trial to Evaluate the Efficacy and Safety of HRS-1893 Tablets in the Treatment of Obstructive Hypertrophic Cardiomyopathy
Brief Title: A Phase III Trial of HRS-1893 in Patients With Obstructive Hypertrophic Cardiomyopathy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS-1893-301
Record Dates: First submitted 2025-06-06; First posted 2025-06-15 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Obstructive Hypertrophic Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HRS-1893 Group (Experimental)
  Interventions: Drug: HRS-1893 Tablets
- HRS-1893 Placebo Group (Placebo Comparator)
  Interventions: Drug: HRS-1893 Placebo Tablets

INTERVENTIONS:
Drug: HRS-1893 Tablets — HRS-1893 tablets.
  Arms: HRS-1893 Group
Drug: HRS-1893 Placebo Tablets — HRS-1893 placebo tablets.
  Arms: HRS-1893 Placebo Group

SUMMARY:
The study is being conducted to evaluate the efficacy and safety of HRS-1893 for obstructive hypertrophic cardiomyopathy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-85 years old, gender unlimited.
2. BMI<35 kg/m2.
3. The diagnosis was obstructive hypertrophic cardiomyopathy.
4. Laboratory determination of echocardiography showed that Rest LVOT-G≥50 mmHg, or Rest LVOT-G≥30 mmHg and LVOT-G≥50 mmHg after Valsalva action.
5. Echocardiographic laboratory tests showed LVEF≥60%.
6. NYHA classification: Grade II - III.
7. Understand the study procedure and sign the informed consent in person, willing to strictly follow the clinical study protocol to complete the study.

Exclusion Criteria:

1. Known or suspected invasive, genetic or storage diseases (e.g. Noonan syndrome, Fabre's disease, amyloidosis) that cause cardiac hypertrophy (similar to oHCM).
2. Had a history of severe valvular heart disease.
3. Abnormal laboratory test results during screening, or any other clinically significant abnormal screening laboratory values, which are determined by the researcher to be unsuitable for inclusion.
4. Other circumstances where the researchers consider the subjects unsuitable to participate in this trial, such as physical or mental illnesses or conditions that may increase the risk of the trial, affect the subjects' compliance with the protocol, or affect the subjects' completion of the trial.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2025-08-11 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
The clinical response rate of treatment with HRS-1893. | After 24 weeks of HRS-1893 treatment.

SECONDARY OUTCOMES:
The incidence of major adverse cardiac events (cardiovascular death, cardiac arrest, non-fatal stroke, non-fatal myocardial infarction, hospitalization for cardiovascular events). | About 29 weeks.
Incidence and severity of any adverse events. | About 29 weeks.
The change in Kansas City Cardiomyopathy Questionnaire - Clinical Summary Score (KCCQ-CSS) from the baseline. | Week 12 and Week 24.

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided